CLINICAL TRIAL: NCT05937685
Title: BP-REACH: Blood Pressure Disparities Reduction, Equity, and Access Among Safety Net Patients With Cardiovascular Health Risk
Brief Title: Reducing Blood Pressure in Patients With High Cardiovascular Risk
Acronym: BP-REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Amytis Towfighi, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1P50MD017366-01 (NIH)
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Infarction; Hypertension; Stroke
Keywords: stroke; myocardial infarction; hypertension; self-management; chronic disease
MeSH Terms: conditions — Myocardial Infarction; Hypertension; Stroke; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants receive the usual care received by patients of the medical center
- Intervention (Experimental): Participants follow the intervention protocol, including receiving educational materials, a home blood pressure monitor, coaching calls from BP REACH coaches and medication management from a pharmacist.
  Interventions: Behavioral: BP REACH Intervention

INTERVENTIONS:
Behavioral: BP REACH Intervention — Educational materials, written and digital. Home blood pressure monitor and self management education from BP REACH coach. Monthly coaching calls from BP REACH coach. Medication management by pharmacist
  Arms: Intervention

SUMMARY:
BP-REACH is a study of a team-based (pharmacist and health coach) program for lowering blood pressure for people with a prior stroke or heart attack in the Los Angeles Department of Health Services healthcare system.

The goal of this clinical trial is to test if this team based program is better at helping people reduce their blood pressure than usual care for people with prior heart attack or stroke. The main questions it aims to answer are:

* Do people in the REACH BP program have lower blood pressure at 12 months compared to those getting usual care?
* Do people in the REACH BP program have better Life's Essential 8 scores and patient experience compared to those getting usual care?

DETAILED DESCRIPTION:
Hypertension is the leading contributor to preventable death and a major risk factor for recurrent cardiovascular events. To enhance BP control after stroke or myocardial infarction (MI), multilevel interventions are needed that incorporate health system and patient level factors.

BP-REACH aims to test the impact of an intervention on systolic blood pressure (SBP) for individuals with a history of stroke or MI in a randomized controlled trial in the Los Angeles Department of Health Services healthcare system. The primary outcome will be change in systolic blood pressure (SBP) at 12 months.

Hypothesis: Patients randomized to the intervention will achieve >2.4 mm Hg greater reduction in SBP at 1 year versus those randomized to usual care.

The study population will include participants from the inpatient and outpatient settings in Los Angeles County Department of Health Services health centers. The participants will be randomized in a 1:1 fashion to usual care or intervention, stratified by site, language and cardiovascular event (myocardial infarction, stroke). Outcomes will be collected from all participants at Baseline, 3 month and 12 month timepoints. The primary outcome is SBP.

Participants randomized to the intervention arm will receive additional a home blood pressure monitor, monthly phone calls from a health coach, and medication initiation and titration by a clinical pharmacist. The pharmacist will follow Los Angeles County Department of Health Services expected practices, which align with the ACC/AHA guidelines for blood pressure control and AHA guidelines for Secondary Stroke Prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients of LA General Medical Center, Rancho Los Amigos, Olive Medical Center or Harbor-UCLA Medical Center with ischemic stroke, hemorrhagic stroke, or myocardial infarction
* English or Spanish speaking
* Systolic blood pressure (SBP) ≥ 130 mm Hg

Exclusion Criteria:

* Age < 35 years
* SBP < 130 mm Hg
* Only speaks a language other than English or Spanish
* Cannot provide informed consent due to dementia or aphasia

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) mmHG | 12 months
  Collected by study staff using blood pressure monitor

SECONDARY OUTCOMES:
Life's Essential 8 | 12 months
  American Heart Association - survey measure. Score of 0-100, with 100 indicating a perfect score for cardiovascular health
BMI (body mass index) | 12 months
  Height (cm) and weight (kg) collected by study staff, height divided by height indicating percentage of fat on the body
Total cholesterol | 12 months
  Lab collection by study staff
HgbA1c (hemoglobin A1C) | 12 months
  Lab collection by study staff
Diet | 12 months
  Survey - California Health Interview Survey
Physical activities | 12 months
  Survey - Behavioral Risk Factor Surveillance System Survey Questionnaire
Smoking | 12 months
  Survey - PATH wave 1 survey

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Casillas, MD, Principal Investigator — University of California, Los Angeles; Amytis Towfighi, MD, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - LA General Medical Center, Los Angeles, California
  - Olive View Medical Center, Sylmar, California
  - Harbor UCLA Medical Center, Torrance, California

IPD SHARING:
Plan to Share IPD: No